CLINICAL TRIAL: NCT02866578
Title: Open Lung Protective Ventilation During Cardiac Surgery With Cardiopulmonary Bypass : a Randomized Controlled Trial
Brief Title: Open Lung Protective Ventilation in Cardiac Surgery
Acronym: PROVECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-03; 2016-A00352-49 (Other: IDRCB)
Record Dates: First submitted 2016-07-07; First posted 2016-08-15 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2016-12

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open lung protective ventilation (Experimental): * Recruitment maneuvers (30 cmH2O during 30 seconds) after intubation, after CPB initiation, before aortic declamping and at ICU arrival.
  * PEEP at 8 cmH2O.
  * Ultraprotective ventilation during CPB: PEEP 8 cmH2O, Tidal volume 3mL/kg, Respiratory rate 12 cycles per minute, FiO2 40%.
  * Assigned intervention - Procedure: patients are randomized and ventilated with the open lung strategy from intubation to detubation.
  Interventions: Procedure: Open lung protective ventilation strategy
- Conventional strategy (No Intervention): No recruitment maneuvers. PEEP at 2 cmH2O. During CPB: continuous positive pressure at 2 cmH2O.

INTERVENTIONS:
Procedure: Open lung protective ventilation strategy
  Arms: Open lung protective ventilation

SUMMARY:
Cardiac surgery with cardiopulmonary bypass (CPB) frequently induces post-operative respiratory dysfunction. The post-operative pulmonary complications (PPCs) significantly increase the peri-operative morbidity and require invasive treatments during longer and more expensive ICU stays. A specific pathophysiology involving general anesthesia and CPB-related factors (inflammation, pulmonary ischemia) has been clearly demonstrated and pulmonary atelectasis seems to play a central role in the occurence of these PPCs. The open lung approach is a ventilation strategy that aims to "open the lung and keep it open" using different ventilatory settings. The efficacy of that strategy is not demonstrated in the global surgical population. However, its application in the perioperative care of cardiac surgery patients could be of great interest by counteracting the development of atelectasis.

The purpose of this multicentre, double blinded, randomized controlled study is to evaluate the influence of a perioperative multimodal protective ventilation strategy based on the "open lung approach" on postoperative outcomes during the first 7 days following cardiac surgery. Participating centres will include 500 adult patients undergoing scheduled on-pump cardiac surgery. The open lung approach will combine recruitment maneuvers (RM), positive end expiratory pressure (PEEP) at 8 cmH2O from intubation to detubation and continuation of ultraprotective ventilation during CPB. It will be compared to a conventional approach without RM, with PEEP at 2 cmH2O and discontinuation of ventilation during CPB. The primary endpoint is any post-operative pulmonary complication. The secondary endpoints are any post-operative extra-pulmonary complications and the number of ICU-free days to day 7.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery planned with CPB and sternotomy.
* Age > 18 years old.

Exclusion Criteria:

* Urgent surgery : cardiac transplantation, aortic dissection, active endocarditis.
* Aortic arch surgery with circulatory arrest.
* LVAD surgery.
* Acute or chronic preoperative hypoxemia (PaO2 < 65 mmHg in air).
* Preoperative shock state requiring catecholamines.
* LVEF < 40%.
* Pulmonary hypertension with systolic pulmonary artery pressure > 50 mmHg.
* Severe right ventricular dysfunction (TDI tricuspid annular systolic velocity < 10 cm.s-1).
* Chronic kidney disease (Glomerular filtration rate < 30 mL/min).
* Body Mass Index > 35kg/m2.
* Patient's refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Post-operative pulmonary complications defined as a composite endpoint | first 7 days post-operatively.
  Mild hypoxemia Moderate hypoxemia Severe hypoxemia Severe bronchospam Radiological atelectasis Respiratory acidosis Pneumonia Pleural effusion Acute Respiratory Distress Syndrome Need for reintubation Need for reintubation

SECONDARY OUTCOMES:
Postoperative extrapulmonary complication | First 7 days post operatively
  Systemic inflammatory response syndrome Sepsis Septic chock Mediastinitis Pericardial tamponade Surgical bleeding Acute kidney failure (KDIGO stage 2 or 3) Postoperative atrial fibrillation Cardiogenic chock Delirium
ICU free Days | First 7 days post operatively
  Days alive and free from the need of intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — AP-HM
Locations (6):
- France (6):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Louis Pradel HCL, Lyon
  - Assistance Publique Hopitaux de Marseille, Marseille
  - CHU MontpellierHôpital Arnaud de VILLENEUVE, Montpellier
  - Hôpital Européen Georges Pompidou AP-HP, Paris
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lagier D, Fischer F, Fornier W, Huynh TM, Cholley B, Guinard B, Heger B, Quintana G, Villacorta J, Gaillat F, Gomert R, Degirmenci S, Colson P, Lalande M, Benkouiten S, Minh TH, Pozzi M, Collart F, Latremouille C, Vidal Melo MF, Velly LJ, Jaber S, Fellahi JL, Baumstarck K, Guidon C; PROVECS Study Group. Effect of open-lung vs conventional perioperative ventilation strategies on postoperative pulmonary complications after on-pump cardiac surgery: the PROVECS randomized clinical trial. Intensive Care Med. 2019 Oct;45(10):1401-1412. doi: 10.1007/s00134-019-05741-8. Epub 2019 Oct 1. PMID 31576435
- [Derived] Lagier D, Fischer F, Fornier W, Fellahi JL, Colson P, Cholley B, Jaber S, Baumstarck K, Guidon C; PROVECS investigators and the ARCOTHOVA group. A perioperative surgeon-controlled open-lung approach versus conventional protective ventilation with low positive end-expiratory pressure in cardiac surgery with cardiopulmonary bypass (PROVECS): study protocol for a randomized controlled trial. Trials. 2018 Nov 13;19(1):624. doi: 10.1186/s13063-018-2967-y. PMID 30424770